CLINICAL TRIAL: NCT04151615
Title: A Multi-center,Open, Longitudinal, Observational Study to Evaluate the Treatment Effectiveness and Safety of the Bortezomib-melphalan-prednisolone Regimen in Treatment-naïve Patients With Multiple Myeloma, Ineligible for Hematopoietic Transplantation
Brief Title: VMP Regimen - Safety, Efficacy, and Optimal Dose Finding Study for Patients With Multiple Myeloma
Acronym: VISION
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-BTZ-OS-401
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Treatment-naïve patients with multiple myeloma who are ineligible for hematopoietic transplantation

SUMMARY:
The 3-drug therapy of Bortezomib-Melphalan-Prednisolone (VMP) is a standard therapy that is commonly used currently in South Korea as a first-line treatment for treatment-naïve patients with multiple myeloma who are ineligible for hematopoietic transplantation. Despite the fact that VMP therapy is outstanding in terms of cost-effectiveness, treatment discontinuation rates due to adverse drug reactions is high. In addition, when considering that the percentage of elderly patients aged 70 years or above in the target patient group is 20% or above, there have been attempts to devise a plan that can decrease side effects while maintaining effectiveness. For example, there have been previous reported cases of overseas applications of modified VMP therapies with reduced doses, but they have applied various combinations in terms of the total cycles, administration intervals, doses, etc. This study was planned to evaluate the overall safety and efficacy of VMP therapy by following up on the actual VMP therapies applied in domestic clinics, patient characteristics, side effect occurrences, administration discontinuation rates, survival data, etc., as well as to collect exploratory data for a more effective study of modified VMP therapies.

This study was planned to evaluate the overall safety and efficacy of VMP therapy by following up on the actual VMP therapies applied in domestic clinics, patient characteristics, side effect occurrences, administration discontinuation rates, survival data, etc., as well as to collect exploratory data for a more effective study of modified VMP therapies.

DETAILED DESCRIPTION:
The data produced when subjects visit the hospital for treatment are collected in case report forms. The follow-up time specified in the following refer to the data collection time. That is, a subject's visit schedule is freely determined by the investigator based on the medical condition of the subject regardless of the follow-up time specified in this protocol, but data that are determined necessary in relation to the study among the data produced during the study period may be collected in CRFs.

In regard to various tests for monitoring of treatment effects including laboratory tests, the corresponding tests are not performed separately for this clinical study, and only those items with existing test results are collected. The following data are collected in CRFs during the study period.

* Demographic information of subjects
* Information on multiple myeloma disease (diagnosis date, diagnosis criteria and related test results, disease stage [ISS and revised ISS], number of osseous lesions)
* Intercurrent diseases
* Height and body weight
* ECOG PS
* IMWG Frailty score
* Laboratory results
* Radiologic results
* Bone marrow examination results
* Supportive therapy administered for symptoms related to multiple myeloma (drug / surgery / radiotherapy)
* Detailed information of administered VMP therapy
* Maintenance therapy / VMP replacement therapy
* Clinical response
* Survival
* Adverse drug reactions related to VMP therapy
* Serious adverse events/adverse drug reactions

ELIGIBILITY:
Inclusion Criteria:

* Patients who provide written consent on the informed consent form for use of personal information after listening to an explanation regarding the purpose, method, etc., of this clinical study
* Adult males and females aged 19 years or above
* Patients without previous experience of treatment for multiple myeloma who have been evaluated as ineligible for hematopoietic transplantation
* Patients scheduled to receive the 3-drug combination (VMP therapy) treatment
* Patients with expected survival period of 6 months or more
* Patients evaluated as having performance status score (ECOG PS) ≤2 (score of 0, 1, 2)
* Patients who have received the following tests within 6 months prior to enrollment

  * Beta2-microglobulin
  * Serum albumin
  * Serum LDH
  * Patients with confirmed del (17), t (4;14), t (14;16) by hybridization FISH test

Exclusion Criteria:

* Patients who have been newly diagnosed with other primary cancers within the last 5 years that can affect the treatment or prognosis of multiple myeloma
* Pregnant women and breast-feeding women
* Patients who are currently participating in other clinical studies (drug or medical device clinical studies) or planning to participate in other clinical studies during the study participation period
* Patients who are determined ineligible to participate in the study by other judgments of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naïve patients with multiple myeloma who are ineligible for hematopoietic transplantation
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
PFS (progression-free survival) | 18 Month after VMP therapy administration
  the survival rate curve of PFS and the median, as well as the 95% confidence interval for this are presented. An event is 'confirmation of progressive disease (PD)' or 'death,' and others are processed as censored at the later time point between the final follow-up time point and the time point of final clinical response evaluation.

SECONDARY OUTCOMES:
ORR (Overall Response Rate) | 18 Month after VMP therapy administration
  The frequency and percentage of subjects who reach CR, VGPR, and PR even once after VMP therapy administration are calculated, and the 95% CI for the percentage is presented.
CR (Complete Response) | 18 Month after VMP therapy administration
  The frequency and percentage of subjects who reach CR even once after VMP therapy administration are calculated, and the 95% CI for the percentage is presented
Time to Response (TTR) | 18 Month after VMP therapy administration
  time to first response and time to best response; here, response must be higher than partial response (PR).
Time to Progression (TTP) | 18 Month after VMP therapy administration
  'confirmation of progressive disease,' and others are processed as censored at the final follow-up time point or the time point of final clinical response evaluation.
Time to Next Treatment (TTNT) | 18 Month after VMP therapy administration
  'administration of VMP replacement therapy (regardless of VMP therapy termination),' and others are processed as censored at the final follow-up
OS (Overall Survival) | 18 Month after VMP therapy administration
  'death,' and others are processed as censored at the final time point with confirmed survival.
Percentage of IMWG frailty scores at Cycle 5 and Cycle 9 | 18 Month after VMP therapy administration
  The frequency and percentage of IMWG frailty scores (Fit: 0 points, Intermediate-fitness: 1 point, Frail: ≥2 points) per time point are presented. The mean, standard deviation, median, minimum value, and maximum value for the variance of IMWG frailty scores at VMP therapy Cycle 5 and Cycle 9 compared to the baseline are summarized with descriptive statistics
Prognosis prediction factors | 18 Month after VMP therapy administration
  * Prognosis variables: PFS/TTR/TTP/OS
  * Potential prediction factors: Age / ISS stage / revised ISS stage / number of osseous lesions / IMWG frailty score at baseline (0 points, 1 point, ≥2 points) / VMP administration pattern

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Jae Kim, Study Director — Boryung Pharmaceutical Co., Ltd
Locations (24):
- South Korea (24):
  - Soonchunhyang University Bucheon hospital, Bucheon-si
  - Inje university Haeundae Paik Hospital, Busan
  - Kosin University Gospel hospital, Busan
  - Pusan national University Hospital, Busan
  - Keimyung University Hospital(Dongsan Medical Center), Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang
  - Gyeongsang National University Changwon Hospital, Gyeongsang
  - Chonnam National University Hwasun Hospital, Hwasun
  - Gachon University Gil Medical Center, Incheon
  - Chungbuk national university Hospital, Jungbuk
  - Dankook University Hospital, Jungnam
  - Chung-Ang University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Ajou University Medical Center, Suwon
  - Ulsan University hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju